CLINICAL TRIAL: NCT00103181
Title: A Randomized Phase III Study of Conventional Whole Breast Irradiation (WBI) Versus Partial Breast Irradiation (PBI) for Women With Stage 0, I, or II Breast Cancer
Brief Title: Radiation Therapy (WBI Versus PBI) in Treating Women Who Have Undergone Surgery For Ductal Carcinoma In Situ or Stage I or Stage II Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Radiation Therapy Oncology Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-39/RTOG 0413; NSABP-B-39; RTOG-0413; SWOG-NSABP-B-39; NCI-2009-00698 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; ductal breast carcinoma in situ; breast cancer in situ; stage IA breast cancer; stage IB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: WBI (Active Comparator): Patients undergo whole breast irradiation (WBI) once daily, 5 days a week for 5-7 weeks.
  Interventions: Radiation: whole breast irradiation
- Group 2: PBI (Experimental): Patients undergo partial-breast irradiation (PBI) twice daily on 5 days over a period of 5-10 days. This may be delivered by intracavitary brachytherapy, MammoSite or other single-entry intracavitary device, or 3-dimensional conformal accelerated partial breast irradiation.
  Interventions: Radiation: 3-dimensional conformal accelerated partial breast irradiation; Radiation: brachytherapy; Radiation: MammoSite or other single-entry intracavitary device

INTERVENTIONS:
Radiation: 3-dimensional conformal accelerated partial breast irradiation
  Arms: Group 2: PBI
Radiation: brachytherapy
  Arms: Group 2: PBI
Radiation: whole breast irradiation — Patients undergo radiation therapy once daily (days 1-5) for up to 7 weeks
  Arms: Group 1: WBI
Radiation: MammoSite or other single-entry intracavitary device
  Arms: Group 2: PBI

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy in different ways may kill any tumor cells that remain after surgery. It is not yet known whether whole breast radiation therapy is more effective than partial breast radiation therapy in treating breast cancer.

PURPOSE: This randomized phase III trial is studying whole breast radiation therapy to see how well it works compared to partial breast radiation therapy in treating women who have undergone surgery for ductal carcinoma in situ or stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare local tumor control in women with ductal carcinoma in situ or stage I or II breast cancer treated with adjuvant whole breast vs partial breast irradiation following lumpectomy.

Secondary

* Compare overall survival, recurrence-free survival, and distant disease-free survival in patients treated with these regimens.
* Compare the cosmetic result in patients treated with these regimens.
* Compare fatigue and treatment-related symptoms in patients treated with these regimens.
* Compare perceived convenience of care in patients treated with these regimens.
* Compare acute and late toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (ductal carcinoma in situ [DCIS] only vs invasive and node negative vs invasive with 1-3 positive nodes), menopausal status (premenopausal vs postmenopausal), hormone receptor status (estrogen receptor [ER]-positive and/or progesterone receptor [PR]-positive vs ER-negative and PR-negative), intention to receive chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms. (Patients who are 50 years of age and over with DCIS regardless of hormone receptor status AND patients with invasive breast cancer meeting all of the following criteria: ≥ 50 years of age, node-negative, and hormone-receptor positive status will not be enrolled in study after 12/30/2006.)

* Group 1: Patients undergo whole-breast irradiation (WBI) once daily, 5 days a week, for 5-7 weeks.
* Group 2: Patients undergo partial-breast irradiation (PBI) twice daily on 5 days over a period of 5-10 days. This may be delivered by multi-catheter brachytherapy, single-entry intracavitary brachytherapy, or 3-D conformal radiotherapy.

Patients in both arms may receive adjuvant chemotherapy at least 2 weeks prior to initiation of WBI OR at least 2 weeks after completion of PBI at the discretion of the treating physician. Patients with ER-positive or PR-positive tumors may also receive hormonal therapy, beginning 3-12 weeks after completion of adjuvant chemotherapy (or before, during, or after completion of WBI or PBI for patients not receiving adjuvant chemotherapy) and continuing for at least 5 years.

After completion of study treatment, patients are followed at 1 and 6 months, every 6 months for 4.5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 4,300 patients (2,150 per treatment arm) will be accrued for this study within 4.6 years. Note: Accrual closed on April 16, 2013, following approval of the Data Monitoring Committee to reduce the sample size from 4,300 to 4,214 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ (DCIS*) or invasive* adenocarcinoma of the breast

  * Stage 0, I, or II disease

    * Stage II tumors must be ≤ 3 cm
  * Gross disease must be unifocal

    * Microscopic multifocality allowed provided total pathological tumor size is ≤ 3 cm
  * No proven multicentric carcinoma in more than 1 quadrant or separated by ≥ 4 cm
  * No non-epithelial breast malignancies (e.g., sarcoma or lymphoma) NOTE: *Patients who are 50 years of age and over with DCIS regardless of hormone receptor status AND patients with invasive breast cancer meeting all of the following criteria: ≥ 50 years of age, node-negative, and hormone-receptor positive status will not be enrolled in study after 12/30/2006
* Prior axillary staging required for patients with invasive breast cancer, including 1 of the following:

  * Sentinel node biopsy alone (if sentinel node is negative)
  * Sentinel node biopsy followed by axillary dissection or sampling with ≥ 6 axillary nodes (if sentinel node is positive)
  * Axillary dissection alone with ≥ 6 axillary nodes
* No more than 3 positive axillary nodes

  * No axillary nodes with definite evidence of microscopic or macroscopic extracapsular extension
  * No positive non-axillary sentinel nodes (intramammary nodes are staged as axillary nodes)
  * No palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes unless there is histologic confirmation that these nodes are negative for tumor
* Must have undergone lumpectomy

  * Resected margins histologically free of tumor
  * Re-excision of surgical margins allowed
  * Target lumpectomy cavity clearly delineated AND target lumpectomy/whole breast reference volume ≤ 30% based on postoperative pre-randomization CT scan
  * Final surgery (i.e., lumpectomy, re-excision of margins, or axillary staging procedure) within the past 42 days
* No suspicious microcalcifications, densities, or palpable abnormalities in the ipsilateral or contralateral breast unless biopsied and found to be benign
* No Paget's disease of the nipple
* No history of invasive breast cancer or DCIS

  * Prior lobular carcinoma in situ treated by surgery alone allowed
* No synchronous bilateral invasive or non-invasive breast cancer
* Partial breast irradiation deemed technically deliverable by radiation oncologist at a credentialed facility
* Must have undergone a history and physical exam within the past 4 months AND a bilateral mammogram within the past 6 months
* Hormone receptor status:

  * Estrogen receptor (ER) status known
  * Progesterone status known if ER analysis is negative
  * Marginal or borderline results are considered positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Premenopausal or postmenopausal

Performance status

* Not specified

Life expectancy

* At least 10 years, excluding diagnosis of breast cancer

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception
* No other malignancy within the past 5 years except previously treated carcinoma in situ of the cervix or colon, melanoma in situ, or basal cell or squamous cell skin cancer

  * Deemed to be at low risk for recurrence
* No collagen vascular disease (e.g., systemic lupus erythematosus or scleroderma), specifically dermatomyositis with a creatine phosphokinase (CPK) level above normal, or active skin rash
* No psychiatric or addictive disorder that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for this malignancy

Chemotherapy

* No prior chemotherapy for this malignancy
* No concurrent chemotherapy during study radiotherapy

Endocrine therapy

* No prior hormonal therapy for this malignancy unless total duration of hormonal therapy was no more than 28 days before randomization
* Concurrent hormonal therapy allowed provided it is not administered during chemotherapy
* No concurrent raloxifene, tamoxifen, or other selective estrogen receptor modulating drugs
* No concurrent hormone replacement therapy
* No concurrent Femring^®

Radiotherapy

* No prior radiotherapy for this malignancy
* No prior breast or thoracic radiotherapy
* No concurrent brachytherapy boosts
* No concurrent intensity modulated radiotherapy
* No concurrent regional nodal irradiation

Surgery

* See Disease Characteristics
* No prior breast implants

  * Patients who have had implants removed are eligible

Other

* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4216 (Actual)
Dates: Start 2005-03; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
In-breast tumor recurrence (IBTR) | every 6 months for 5 years; annually thereafter for up to 10 years

SECONDARY OUTCOMES:
Overall survival | time from randomization to death due to any cause assessed up to 15 years
Recurrence-free survival | time from randomization to recurrence assessed every 6 months for 5 years and annually thereafter for up to 10 years
Distant disease-free survival | time from randomization to event occurrence assessed every 6 months for 5 years and annually thereafter for up to 10 years
Quality of life and patient-reported cosmesis by Breast Cancer Treatment Outcome Scale, MOS SF-36 Vitality, Convenience of Care scale, and symptoms | measured at baseline, and 1 and 6 months and 1, 2, and 3 years after completion of study treatment
Toxicity as assessed by adverse events during treatment | at end of RT, and 4 weeks, 6 months, 12 months; every 6 months for years 2 through 5; and annually thereafter for up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (387):
- United States (374):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Arizona Breast Cancer Specialists, Scottsdale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Auburn Radiation Oncology, Auburn, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - North Bay Cancer Center, Fairfield, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Community Hospital of the Monterey Peninsula Comprehensive Cancer Center, Monterey, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Feather River Hospital Cancer Center, Paradise, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Mercy Regional Cancer Center at Mercy Medical Center, Redding, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Sharp Memorial Hospital Cancer Center, San Diego, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Stanford Cancer Center, Stanford, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Ruby L. Golleher Cancer Program at Presbyterian Intercommunity Hospital, Whittier, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Connecticut Oncology & Hematology - Torrington, Torrington, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Kootenai Cancer Center - Coeur d'Alene, Coeur d'Alene, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Good Samaritan Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Illinois CancerCare - Cottage, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - CCOP - Kansas City, Prairie Village, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - NSMC Cancer Center - Peabody, Danvers, Massachusetts
  - MetroWest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Payson Center for Cancer Care at Concord Hospital, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Memorial Sloan-Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - Trinitas Comprehensive Cancer Center at Trinitas Hospital, Elizabeth, New Jersey
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - St. Francis Regional Cancer Center, Trenton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Cayuga Medical Center of Ithaca, Ithaca, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Saint Francis Hospital Cancer Center, Poughkeepsie, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Cancer Centers of North Carolina - Raleigh, Raleigh, North Carolina
  - Coastal Carolina Radiation Oncology Center, Wilmington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Intercommunity Cancer Center, Monroeville, Pennsylvania
  - Norristown Regional Cancer Center, Norristown, Pennsylvania
  - Drexel University College of Medicine - Center City Hahnemann Campus, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Northmain Radiation Oncology, Providence, Rhode Island
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Georgetown Memorial Hospital, Georgetown, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center - Denton South, Denton, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor Medical Center at Irving, Irving, Texas
  - Texas Oncology, PA at Lake Vista Cancer Center, Lewisville, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology, PA at Texas Cancer Center Round Rock, Round Rock, Texas
  - Cancer Care Centers of South Texas - Northeast, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
- Canada (11):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- University College Hospital, Galway, Ireland
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Croshaw R, Kim Y, Lappinen E, Julian T, Trombetta M. Avoiding mastectomy: accelerated partial breast irradiation for breast cancer patients with pacemakers or defibrillators. Ann Surg Oncol. 2011 Nov;18(12):3500-5. doi: 10.1245/s10434-011-1784-2. Epub 2011 May 24. PMID 21607774
- [Background] Hasan Y, Kim L, Wloch J, Chi Y, Liang J, Martinez A, Yan D, Vicini F. Comparison of planned versus actual dose delivered for external beam accelerated partial breast irradiation using cone-beam CT and deformable registration. Int J Radiat Oncol Biol Phys. 2011 Aug 1;80(5):1473-6. doi: 10.1016/j.ijrobp.2010.04.013. Epub 2010 Jul 23. PMID 20656415
- [Background] Hepel JT, Tokita M, MacAusland SG, Evans SB, Hiatt JR, Price LL, DiPetrillo T, Wazer DE. Toxicity of three-dimensional conformal radiotherapy for accelerated partial breast irradiation. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1290-6. doi: 10.1016/j.ijrobp.2009.01.009. Epub 2009 Apr 22. PMID 19395195
- [Background] Kainz K, White J, Herman J, Li XA. Investigation of helical tomotherapy for partial-breast irradiation of prone-positioned patients. Int J Radiat Oncol Biol Phys. 2009 May 1;74(1):275-82. doi: 10.1016/j.ijrobp.2008.11.028. PMID 19362247
- [Background] Langen KM, Buchholz DJ, Burch DR, Burkavage R, Limaye AU, Meeks SL, Kupelian PA, Ruchala KJ, Haimerl J, Henderson D, Olivera GH. Investigation of accelerated partial breast patient alignment and treatment with helical tomotherapy unit. Int J Radiat Oncol Biol Phys. 2008 Mar 15;70(4):1272-80. doi: 10.1016/j.ijrobp.2007.11.019. Epub 2008 Jan 22. PMID 18207666
- [Background] Wojcicka JB, Lasher DE, Malcom R, Fortier G. Clinical and dosimetric experience with MammoSite-based brachytherapy under the RTOG 0413 protocol. J Appl Clin Med Phys. 2007 Oct 24;8(4):176-184. doi: 10.1120/jacmp.v8i4.2654. PMID 18449152
- [Background] Akbari M, Russo SA, Jacobson JS, et al.: Association of women's local treatment decisions with local recurrence risk and life expectancy. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2035, S228-9, 2006.
- [Background] Burch D, Langen KM, Buchholz D, et al.: Partial breast irradiation with helical tomotherapy using RTOG 0413 planning constraints. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2047, S235-6, 2006.
- [Background] Hiatt JR, Evans SB, Price LL, Cardarelli GA, Dipetrillo TA, Wazer DE. Dose-modeling study to compare external beam techniques from protocol NSABP B-39/RTOG 0413 for patients with highly unfavorable cardiac anatomy. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1368-74. doi: 10.1016/j.ijrobp.2006.03.060. PMID 16863924
- [Background] Bovi JA, Li XA, White J, et al.: Comparison of three partial breast irradiation techniques: treatment effectiveness based upon biological models. [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A-1061, S181, 2005.
- [Background] Dickler A. The MammoSite breast brachytherapy device: targeted delivery of breast brachytherapy. Future Oncol. 2005 Dec;1(6):799-804. doi: 10.2217/14796694.1.6.799. PMID 16556059
- [Background] Sanghani M, Wazer DE. Patient selection for NSABP B-39/RTOG 0413: have we posed the right questions in the right way? Brachytherapy. 2007 Apr-Jun;6(2):119-22. doi: 10.1016/j.brachy.2007.01.002. No abstract available. PMID 17434104
- [Result] Julian TB, Costantino JP, Vicini FA, et al.: Early toxicity results with 3D conformal external beam therapy (CEBT) from the NSABP B-39/RTOG 0413 accelerated partial breast irradiation (APBI) trial. [Abstract] J Clin Oncol 29 (Suppl 15): A-1011, 2011.
- [Result] Jain AK, Vallow LA, Gale AA, Buskirk SJ. Does three-dimensional external beam partial breast irradiation spare lung tissue compared with standard whole breast irradiation? Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):82-8. doi: 10.1016/j.ijrobp.2008.10.041. Epub 2009 Feb 21. PMID 19231103
- [Result] Tendulkar RD, Chellman-Jeffers M, Rybicki LA, Rim A, Kotwal A, Macklis R, Obi BB. Preoperative breast magnetic resonance imaging in early breast cancer: implications for partial breast irradiation. Cancer. 2009 Apr 15;115(8):1621-30. doi: 10.1002/cncr.24172. PMID 19224552
- [Result] Patel RR, Christensen ME, Hodge CW, Adkison JB, Das RK. Clinical outcome analysis in "high-risk" versus "low-risk" patients eligible for national surgical adjuvant breast and bowel B-39/radiation therapy oncology group 0413 trial: five-year results. Int J Radiat Oncol Biol Phys. 2008 Mar 15;70(4):970-3. doi: 10.1016/j.ijrobp.2007.12.005. PMID 18313521
- [Result] Al-Hallaq H, Mell L, Advani S, et al.: Magnetic resonance imaging (MRI) identifies multifocal and multicentric disease in breast cancer patients eligible for the NSABP B-39/RTOG 0413 partial breast irradiation (PBI) trial. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1086, S179-S180, 2006.
- [Derived] Ganz PA, Cecchini RS, White JR, Vicini FA, Arthur DW, Rabinovitch RA, Kuske RR, Julian TB, Parda DS, Scheier MF, Winter KA, Paik S, Kuerer HM, Vallow LA, Pierce LJ, Mamounas EP, McCormick B, Bear HD, Germain I, Gustafson GS, Grossheim L, Petersen IA, Hudes RS, Curran WJ Jr, Wolmark N. Quality-of-life outcomes from NRG Oncology NSABP B-39/RTOG 0413: whole-breast irradiation vs accelerated partial-breast irradiation after breast-conserving surgery. J Natl Cancer Inst. 2025 Jan 1;117(1):103-111. doi: 10.1093/jnci/djae219. PMID 39254630
- [Derived] Vicini FA, Cecchini RS, White JR, Arthur DW, Julian TB, Rabinovitch RA, Kuske RR, Ganz PA, Parda DS, Scheier MF, Winter KA, Paik S, Kuerer HM, Vallow LA, Pierce LJ, Mamounas EP, McCormick B, Costantino JP, Bear HD, Germain I, Gustafson G, Grossheim L, Petersen IA, Hudes RS, Curran WJ Jr, Bryant JL, Wolmark N. Long-term primary results of accelerated partial breast irradiation after breast-conserving surgery for early-stage breast cancer: a randomised, phase 3, equivalence trial. Lancet. 2019 Dec 14;394(10215):2155-2164. doi: 10.1016/S0140-6736(19)32514-0. Epub 2019 Dec 5. PMID 31813636